CLINICAL TRIAL: NCT07286994
Title: Randomized-controlled Trial of Remotely-deployed Gamification Interventions to Increase Physical Activity in Veterans With Parkinsons Disease
Brief Title: Gamification and Physical Activity in PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NURM-003-25S
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Exercise; Economics, Behavioral
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Behavior

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to either a gamification intervention or control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gamification (Experimental): Subjects will participate in an automated gamification intervention with loss or gain of points based on reaching a step goal target
  Interventions: Behavioral: Gamification
- Feedback control (Active Comparator): Subjects in the control group will only receive a daily text message reminding them of their daily step goal and whether they met the goal or not
  Interventions: Behavioral: Feedback control

INTERVENTIONS:
Behavioral: Gamification — Subjects will participate in an automated gamification intervention with loss or gain of points based on reaching a step goal target
  Arms: Gamification
Behavioral: Feedback control — Subjects in the control group will only receive a daily text message reminding them of their daily step goal and whether they met the goal or not
  Arms: Feedback control

SUMMARY:
Despite overwhelming evidence that exercise can improve motor and non-motor symptoms of Parkinson's Disease (PD), less than 25% of Veterans with PD meet recommended activity goals. Interventions to increase PA that are scalable and can be deployed in the community represent a major opportunity. The investigators' preliminary work has demonstrated that gamification, a method commonly used for health promotion, can lead to increases in physical activity in PD. In this study, the investigators will test the effectiveness of gamification in a randomized trial to increase activity. Importantly, the investigators will also examine the effect of step count and exercise intensity on clinical outcomes and explore factors important to widespread implementation of the program VA.

DETAILED DESCRIPTION:
Background/Significance: Exercise and physical activity (PA) improve PD symptoms and have been hypothesized to modify disease onset and progression. Further, exercise has been shown to improve debilitating non-motor symptoms (NMS, including depression, sleep, cognition) that are unresponsive or even worsened by dopaminergic treatments used to improve motor symptoms. Most of this evidence comes from resource-intensive, short-term observed trials of exercise, while the investigators' work and that of others has demonstrated low free-living activity levels in PD that worsen with disease duration. In fact, less than 25% of Veterans meet recommended activity goals. Interventions to increase PA that are scalable and can be deployed in the community represent a major opportunity and unmet need in PD. Behavioral economics-based interventions employing wearable devices (i.e. gamification) are well defined and have successfully increased PA in a variety of populations but have not been studied in individuals with chronic neurologic diseases like PD. Such interventions can also be individualized, remotely deployed and scaled widely to increase access. The investigators' preliminary data from an open-label feasibility trial demonstrate that Veterans with PD are: 1) willing and able to adopt technologies required for the intervention; and 2) respond to the intervention, increasing step counts by ~20%.

Innovation: This will be the first randomized clinical trial to incorporate behavioral economic principles using gamification to increase physical activity among Veterans with PD. It will also be innovative by directly examining the impact of these interventions on clinical outcomes rather than just step counts. Further we will investigate the relationship between increasing steps alone compared to exercise intensity and clinical outcomes. To improve scalability and decrease burden on Veterans, the entire study will be conducted completed remotely including enrollment and interventions.

Specific Aims: Aim 1: To determine whether remotely deployed gamification interventions in Veterans with PD improve physical activity PA levels measured by average daily step counts using Fitbits. Aim 2: To determine whether changes in PA resulting from gamification affect motor symptoms in Veterans with PD (tremor, bradykinesia, immobility) measured by wearable sensors (Parkinson's KinetiGraph,PKG). Aim 3: To determine whether changes in PA resulting from gamification interventions affect NMS measured using validated questionnaires completed through a web-based digital health platform. Aim 4: To conduct a qualitative process evaluation and implementation analysis to inform implementation efforts within VA.

Methodology: Veterans with PD (n=110) will be enrolled into a randomized, controlled trial comprised of a 12-week intervention and a 12-week follow-up. Wearable devices will be used to passively monitor physical activity levels (steps and moderate/vigorous, MVPA). Clinical outcomes will be captured by the PKG (motor parkinsonism) and validated questionnaires completed through a digital health platform (non-motor symptoms) Interventions will be deployed using Way to Health, a technology platform that the investigators have demonstrated is feasible to use within the VA Health System. Outcomes will include physical activity in steps (primary), MVPA and motor and non-motor clinical outcomes.

Impact: Personalized strategies using digital health technology to increase physical activity would be highly scalable with broad reach, improving the symptoms and lives of countless people living with PD.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Have a clinical diagnosis of PD based on diagnosis codes and chart review
* Are on a stable regimen of anti-parkinsonian medication

Exclusion Criteria:

* Diagnosis of an atypical parkinsonian syndrome or concomitant administration of a drug that could cause parkinsonian syndromes
* Cardiovascular or other medical comorbidities that preclude participation in an intervention to increase physical activity
* Lack of access to a smartphone or other device (tablet or networked computer) that can be used to interface with the Fitbit app and Way to Health platform
* Fallen more than twice within the past year (assessed via phone screening)
* Clinical diagnosis of dementia

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in step counts | end of intervention period (week 26)
  Primary outcome: change in daily step counts from baseline to intervention. H1a: subjects randomized to gamification will increase step counts significantly more than controls.
Bradykinesia | end of intervention period (week 26)
  Primary outcome: association between changes in step count and changes in bradykinesia. Bradykinesia scores are measured during the last week of the study period using the wrist-worn PKG by Empatica device. Bradykinesia scores are numeric, with higher numbers indicating more severe symptoms.
Non-motor symptoms questionnaire (NMSQ) | end of intervention period (week 26)
  Association between changes in step count and changes in NMSQ during the intervention. The NMSQ is a well-validated 30-item questionnaire assessing the severity of non-motor symptoms in PD. Questions are subdivided into various non-motor domains (cardiovascular, sleep, mood, hallucinations, memory, GI, urinary, sexual function, and miscellaneous). Higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Change in Moderate/Vigorous Physical Activity (MVPA) | end of intervention period (week 26)
  Comparison of changes in MVPA comparing gamification to control subjects. MVPA is measured using the wrist-worn Fitbit device. The Fitbit app calculates an average number of minutes/day in MVPA.

CONTACTS AND LOCATIONS:
Overall Officials: James F Morley, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No